CLINICAL TRIAL: NCT00845988
Title: Metabolic Effects of Switching to Aripiprazole in Patients With Bipolar Disorders Having Drug-induced Weight Gain
Brief Title: Metabolic Effects of Switching to Aripiprazole in Patients With Bipolar Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kyooseob Ha, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-2008-104
Record Dates: First submitted 2009-02-14; First posted 2009-02-18 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Bipolar Disorders; Metabolic Complication
Keywords: Bipolar disorder; metabolic complication; Aripiprazole; Weight gain; Clinical Trial; Antipsychotic; Metabolic syndrome; Psychopharmacology; Open Label
MeSH Terms: conditions — Bipolar Disorder; Weight Gain; Metabolic Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment as usual (Active Comparator): patients showing weight gain while receiving treatment with risperidone, olanzapine, quetiapine, or clozapine
  Interventions: Drug: aripiprazole
- switch to aripiprazole (Experimental): aripiprazole
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: aripiprazole — dosage form : po recommended dosage : more than 10mg/day duration : 28 weeks

SUMMARY:
The primary goal of this study is to investigate metabolic changes and maintaining efficacy in stabilized patients with bipolar disorders who have pharmacologically induced weight gain.

DETAILED DESCRIPTION:
* reduced treatment adherence due to metabolic side effects
* suggested advantages of aripiprazole in metabolic profile over other antipsychotics or mood stabilizers
* randomized trial of switch from previous drugs to aripiprazole

ELIGIBILITY:
Inclusion Criteria:

* patients with bipolar disorders (I, II, NOS) diagnosed with DSM-IV criteria
* age between 18 and 65
* Decisional capacity is adequate to provide informed consent or has an authorized appropriate surrogate decision maker. in a syndromal remission state at least for 2 months : CGI - BP ≤ 3
* patients who have exhibited a clinically significant increase in body weight after starting the administration of their current antipsychotic (ie >7% weight gain)

Exclusion Criteria:

* diagnosis of eating disorder, substance abuse, and psychotic disorder
* history of neurological and medical illness
* pregnant or breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Weight BMI Glucose and lipid profiles CGI-BP KOQOL SWN-K | 0, 4, 8, 12, 18, 26 week

SECONDARY OUTCOMES:
ECG prolactin SAS BAS UKU-SERS-Pat-Korean version | 0, 4, 8, 12, 18, 26 week

CONTACTS AND LOCATIONS:
Overall Officials: Kyooseob Ha, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea